CLINICAL TRIAL: NCT04483167
Title: Phase I Study, Prospective, Monocentric, Uncontrolled, Non-randomized, Open, Interventional. First Human Administration of an Inflammation Tracer (99mTc-cAbVCAM1-5) Using the Scintigraphy in Healthy Volunteers and Asymptomatic Patients.
Brief Title: Clinical Transfer of a Vulnerable Atherosclerotic Plaque Tracer : 99mTc-cAbVCAM1-5 (ATHENA)
Acronym: ATHENA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC19.051
Record Dates: First submitted 2020-03-09; First posted 2020-07-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases; Atherosclerosis
Keywords: 99mTc-cAbVCAM1-5; intravenous injection
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: 7 healthy volunteers (1+3+3) and 6 asymptomatic patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 99mTccAbVCAM1-5 (Experimental): Healthy volunteers and asymptomatic patients
  1. Pré-screening of the volunteers by the CIC or the Vascular Surgeon and sending or handing over the newsletter
  2. Visit 0 Selection: Validation of IC / NIC + Consent collection + additional exams
  3. Visit 1 Inclusion: J0 Scintigraphic imaging following injection 99mTc-cAbVCAM1-5 (370 MBq - 550 MBq - 750 MBq depend of the SAE or AE )
  4. Visit 2: Follow-up visit (Day 14 +/- 7 days post injection)
  5. Visit 3: End of the study, follow-up visit (70 days +/- 10 days post injection)
  Interventions: Drug: 99mTccAbVCAM1-5 injection

INTERVENTIONS:
Drug: 99mTccAbVCAM1-5 injection — intravenous injection of 99mTccAbVCAM1-5 with dose increase

SUMMARY:
Clinical Transfer of a Tracer of the Vulnerable Atheroma Plate: 99mTc-cAbVCAM1-5. (ATHENA).

This is a phase I/IIa, prospective, monocentric, non-controlled, non-randomized, open-label, interventional study.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide with more than 17.6 million deaths. Of these 17.6 millions deaths, 15 millions (85.1%) are attributable to coronary heart disease and cerebrovascular disease, and in both cases the main etiology is atherosclerosis.

In the coronary arteries, while the presence of a stenosing atherosclerotic plate can be detected by the coronary angiography technique that allows visualization of the lumen of the vessels, the same cannot be said of a plate that is vulnerable to eccentric remodeling. Indeed, this plate has little or no effect on the lumen of the artery. As a result, it is undetectable on coronary angiography. These vulnerable coronary atheromatous plaques are characterized by intense inflammatory phenomena leading to the formation of a large lipidic and necrotic heart covered by a thin fibrous capsule. They are prone to rupture, with the immediate consequence of the formation of a thrombus that can cause ischemia and necrosis of the downstream myocardial territory. In practice, 68% of myocardial infarctions are caused by the rupture of vulnerable plaques resulting in stenosis of less than 50% of the vascular lumen. In addition, in two-thirds of cases the infarction is the inaugural clinical event of coronary artery disease.

Currently, there are no validated non-invasive techniques for diagnosing vulnerable atheroma plate. In this context, the Laboratory Radiopharmaceutiques Biocliniques (LRB, UMR_S1039), has selected Vascular Cell Adhesion Molecule 1 (VCAM-1) as a potential target for molecular imaging of vulnerable plate. Indeed, in the arterial tree, its expression is restricted to atheromatous plates presenting an inflammatory phenotype which is considered a major vulnerability criterion. A radiopharmaceutical targeting VCAM-1 (99mTccAbVCAM1-5) has therefore been developed and validated in preclinical studies.

The final objective of this project is to evaluate in clinical practice the potential of this new imaging agent for the non invasive diagnosis of the vulnerable atheroma plates.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Ages 18-55
* No nuclear imaging or CT scans in the year prior to inclusion
* A person not exposed to ionizing radiation according to the labour code.

Patients:

* Ages between 18 and 80
* Atherosclerosis with asymptomatic carotid atheroma plate.
* Indication of carotid endarterectomy.

All:

* Person affiliated with or benefiting from social security
* Person who has given written informed consent

Non inclusion Criteria:

* Woman of childbearing potential in the absence of highly effective contraception or man of childbearing potential without mechanical contraception.
* Medical history that significantly interferes with biodistribution
* History of disease which may impair the absorption, diffusion and excretion of the radiopharmaceutical: Crohn's disease, celiac disease.
* Known allergy to one of the constituents of the product.
* Intoxication with alcohol or drugs on purpose
* Grade 3 haematological toxicity for the following parameters : Hemoglobin, platelets, leukocytes and neutrophil polynuclear cells.
* Grade 2 renal toxicity for the following parameters: Urea and creatinine and/or Glomerular filtration rate according to the CPK-EPI formula < 60mL/min/1.73m².
* Grade 2 liver toxicity for the following parameters : AST, ALT, GGT, PAL and bilirubin.
* Grade 2 pancreatic toxicity for the following parameter: lipase.
* Blood or urine pregnancy test (confirmed in blood) inconclusive or positive for women of childbearing potential.
* Participation in other research involving the type 1 or 2 human being at the same time
* Person in a period of exclusion from other research involving the human person
* Living conditions suggesting an inability to follow all the visits provided for in the protocol.
* Subject who would receive more than 4,500 euros in compensation as a result of participation in other research involving the human person in the 12 months preceding this study.
* Subject not contactable in case of emergency
* Protected person (Sections L1121-5 to L1121-8 of the CSP)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by all adverse event according to the NCI Common Terminology Criteria for Adverse Events (CTCAE)_v5.0_2017-11-27. | 70 days after IP injection +/- 10 days
  All Adverse events reported according to according to the NCI Common Terminology Criteria for Adverse Events (CTCAE)_v5.0_2017-11-27.
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by biological parameters. | 24 hours for healthy volonteers, 6 hours for patients.
  Total Cholesterol (g/L)
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by biological parameters. | 24 hours for healthy volonteers, 6 hours for patients.
  Liver enzymes (ASAT - ALAT - GGT)
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by biological parameters. | 24 hours for healthy volonteers, 6 hours for patients.
  Total bilirubin
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by Electrocardiogram. | 24 hours for healthy volonteers, 6 hours for patients and 14 days after IP injection +/- 7 days + 70 days after IP injection for each group
  ECG (P Wave, QRS Complex, QT Interval)
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by vital signs. | 24 hours for healthy volonteers, 6 hours for patients and 14 days after IP injection +/- 7 days + 70 days after IP injection for each group
  Blood preasure (mmHg)
Evaluation of 99mTc-cAbVCAM1-5 adverse events as assessed by vital signs. | 24 hours for healthy volonteers, 6 hours for patients and 14 days after IP injection +/- 7 days + 70 days after IP injection for each group
  Heart rate (beats/min)

SECONDARY OUTCOMES:
Assessment of biodistribution in all subjects included in the study (healthy volunteers + patients) | 24 hours for healthy volonteers, 6 hours for patients.
  Radioactive activity (MBq) measured in urine, blood and stool + full body images
Dosimetry evaluation of 99mTc-cAbVCAM1-5 in healthy volunteers and patients. | 24 hours for healthy volonteers, 6 hours for patients.
  Dosimetry mesured in healthy subjects and patients in the different organs
Evaluation of the feasibility of the technique using 99mTccAbVCAM1-5 as a tracer for the vulnerable atheroma plate. | 3 hours after injection
  Verification of the concordance between the expression of VCAM-1 in imaging and on operative part of carotid endarterectomy in patients. Comparison between the intensity of the 99mTc-cAbVCAM1-5 signal observed at the level of the carotids and the level of expression of VCAM-1 determined on an operative endarterectomy part of the carotid concerned, by immunohistochemistry and / or ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DE LEIRIS, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116
- [Background] Little WC, Constantinescu M, Applegate RJ, Kutcher MA, Burrows MT, Kahl FR, Santamore WP. Can coronary angiography predict the site of a subsequent myocardial infarction in patients with mild-to-moderate coronary artery disease? Circulation. 1988 Nov;78(5 Pt 1):1157-66. doi: 10.1161/01.cir.78.5.1157. PMID 3180375